CLINICAL TRIAL: NCT00839631
Title: A Phase 1, Open Label, Dose Escalation Study Evaluating the Safety and Pharmacokinetics of Enteric Coated D-3263 Hydrochloride in Subjects With Advanced Solid Tumors
Brief Title: Dose Escalation Study of EC D-3263 HCl in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T08-1
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Solid Tumors
Keywords: subjects with advanced solid tumors refractory to standard therapy or for whom no effective therapy is available.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: EC D-3263 HCl — EC D-3263 HCl, capsules, 50 mg. Oral administration. Dose escalation cohorts (cycle one: single dose on Day 1, daily doses on day 8-28; subsequent cycles: 1 week drug holiday followed by 3 weeks of daily dosing). Expansion Cohort: daily dosing for 28 days followed by a single 7 day drug holiday (Cycle 1), continuing thereafter with daily dosing.

SUMMARY:
This is a Phase 1, dose escalation study evaluating safety and pharmacokinetics of enteric coated D-3263 HCl in subjects with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed advanced solid tumor malignancy which is either refractory to standard therapy or for which no standard therapy exists
* measurable or evaluable disease
* >= 18 years of age
* ECOG of 0, 1 or 2
* no treatement with chemotherapy, radiotherapy or other systemic therapy (excluding depot LHRH agonist or antagonist for subjects with prostate cancer) for the treatment of his or her tumor with in 28 days prior to receipt of EC D-3263 HCl

Exclusion Criteria:

* Clinically significant coronary artery disease or conduction system abnormality
* Coagulation disorder
* Active infection requiring the use of systemic antimicrobial medications within seven days prior to receipt of EC D-3263 HCl
* Any major surgery within 28 days prior to receipt of EC D-3263 HCl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Assess the safety of EC D-3263 HCl | weekly
Determine the maximum tolerated dose of EC D-3263 HCl administered orally daily | weekly

SECONDARY OUTCOMES:
Characterize the pharmacokinetic profile of EC D-3263 HCl after a single dose and repeat daily dosing | periodically within the first month, weekly thereafter
preliminary assessment of antitumor activity | 1 month, periodically thereafter

CONTACTS AND LOCATIONS:
Locations (1):
- South Texas Accelerated Research Therapeutics (START), San Antonio, Texas, United States